CLINICAL TRIAL: NCT00623155
Title: Evaluation of a Malaria Transmission Target Strategy Based on the Periodic Treatment With Sulfadoxine-Pyrimethamine vs. Early Case Management
Brief Title: Seasonal Intermittent Preventive Treatment With Sulfadoxine-Pyrimethamine in Children in Mali
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bamako (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Dr. Alassane Dicko, Faculty of Medicine, Pharmacy and Dentistry, University of Bamako
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A10828
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2008-02-25 (Estimated); Status verified 2002-09

CONDITIONS: Malaria
Keywords: malaria; intermittent preventive treatment; season; children
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Control group
- 2 (Experimental): Test group
  Interventions: Drug: Seasonal IPT in children - Sulfadoxine-pyrimethamine

INTERVENTIONS:
Drug: Seasonal IPT in children - Sulfadoxine-pyrimethamine — Subjecs randomized to receive two intermittent preventive treatments with standard recommended treatment doses of Sulfadoxine-pyrimethamine at 8 weeks interval during the peak malaria transmission season.
  Arms: 2

SUMMARY:
Recent, randomized controlled trials conducted in areas of perennial malaria transmission have shown that intermittent preventive treatment (IPT) given at the time of vaccination reduced the incidence of the first episode of malaria and severe anaemia during the first year of life by more than 50% without there being any rebound in the subsequent year. However, in countries such as Mali, where malaria is highly seasonal and prevalent in older children, IPT in infants may not be the optimum way in which to use antimalarial drugs to prevent malaria. An alternative approach is to give intermittent preventive treatment to children at risk just during the rainy season. Here we propose (i) to evaluate the impact of two seasonal IPT (sIPT) with Sulfadoxine-pyrimethamine (SP) given at 8 weeks interval on the incidence of malaria disease in children of 6 months to 10 years in an area of seasonal transmission, in Kambila, Mali; (ii) to assess the impact of this strategy on the in vivo response of P. falciparum to SP; (iii) to assess the potential rebound effect of this strategy on the subsequent transmission season after the cessation. Children 6 months-10 years in Kambila, Mali will randomized to receive either IPT with SP twice at 8 weeks interval or no IPT during the transmission season and will followed up for 12 months. Subjects will be also followed during the subsequent transmission season to assess possible rebound effect. Clinical malaria cases will be treated with SP and followed for 28 days to assess the in vivo response during both periods.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 10 years
* Agree to seek initial medical care for all medical illness in the study clinic during the study period
* Written informed consent by a parent or legal garden,
* No plan to travel for a long time during the study period.

Exclusion Criteria:

* History of allergy to sulfa drugs or Sulfadoxine-pyrimethamine
* Chronic illness or symptomatic malaria at the time of enrollment

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 262 (Actual)
Dates: Start 2002-07; Primary Completion 2003-07 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
incidence rate of clinical malaria
in vivo adequate clinical and parasitological response of P. falciparum to SP

CONTACTS AND LOCATIONS:
Overall Officials: Ogobara Doumbo, MD, Study Director — University of Bamako; Alassane Dicko, MD, Principal Investigator — University of Bamako
Locations (1):
- Malaria Research and Training Center, Faculty of Medicine Pharmacy and Dentistry, University of Bamako, Bamako, Mali

REFERENCES:
- [Derived] Dicko A, Sagara I, Sissoko MS, Guindo O, Diallo AI, Kone M, Toure OB, Sacko M, Doumbo OK. Impact of intermittent preventive treatment with sulphadoxine-pyrimethamine targeting the transmission season on the incidence of clinical malaria in children in Mali. Malar J. 2008 Jul 8;7:123. doi: 10.1186/1475-2875-7-123. PMID 18611271